CLINICAL TRIAL: NCT00517192
Title: A Prospective, Randomized, Open-labelled, Multi-centre Trial Comparing the Safety and Efficacy of Ritonavir-boosted Aptivus (Tipranavir, TPV/r) to That of Prezista® (Darunavir, DRV/r) in Three-class (NRTI, NNRTI, and PI) Treatment-experienced Patients With Resistance to More Than One PI. POTENT: PrOspecTive EvaluatioN of Tipranavir vs. Darunavir in Treatment Experienced Patients
Brief Title: Comparison of TPV/r to DRV/r in Triple Class Experienced Patient With Resistance to > 1 PI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1182.71
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Results first posted 2009-10-23 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Darunavir; Ritonavir

INTERVENTIONS:
Drug: Tipranavir
Drug: Darunavir
Drug: Ritonavir

SUMMARY:
The objective of this study is to compare the efficacy and safety of Tipranavir/ritonavir (TPV/r, 500mg/200mg twice daily) to the safety and efficacy of Darunavir/ritonavir (DRV/r 600 mg /100 mg twice daily) in combination with investigator selected optimised background regimens in patients who are three-class (Nucleoside reverse transcriptase inhibitors (NRTI), Nonnucleoside reverse transcriptase inhibitors (NNRTI), and Protease inhibitor (PI)) treatment-experienced (a minimum of 3-months duration for each class) with resistance to more than one PI on the screening virtual phenotype resistance testing.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to trial participation.
2. HIV-1 infected male or female >18 years of age.
3. Three-class (NRTI, NNRTI, and PI) treatment-experienced patients (a minimum of 3-months duration for each class or documented class hypersensitivity/intolerance) with resistance (minimal or reduced response) to more than one PI on the screening virtual phenotype resistance testing. In the case of NNRTIs, NNRTI resistance in the absence of exposure is equivalent to being NNRTI treatment experienced.
4. Patient's optimized background regimen must contain one of the following ARV options:

   * A minimum of two genotypically active nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) reported as "maximal response" or "sensitive" on the screening virtual phenotype report.
   * A minimum of one genotypically active NRTI reported as "maximal response" or "sensitive" on the screening virtual phenotype report plus Enfuvirtide if not used previously.
   * A minimum of one genotypically active NRTI reported as "maximal response" or "sensitive" on the screening virtual phenotype report plus an integrase inhibitor if not used previously and if available through an expanded access program and allowed by local regulatory authorities.
   * A minimum of one genotypically active NRTI reported as "maximal response" or "sensitive" on the screening virtual phenotype report plus the CCR5 chemokine receptor antagonist Maraviroc if available through an expanded access program, not used previously and allowed by local regulatory authorities.
   * Zero or one genotypically active NRTI reported as "maximal response" or "sensitive" on the screening virtual phenotype report plus two of the following drugs, Enfuvirtide, an integrase inhibitor and Maraviroc if available, not used previously and allowed by local regulatory authorities.
   * Two genotypically partially active NRTIs (provided that they are not part of the current failing regimen) reported as "reduced response" on the screening virtual phenotype report plus one of the following drugs, Enfuvirtide, an integrase inhibitor or Maraviroc if available, not used previously and allowed by local regulatory authorities.
5. Patient has been on their current (failing) PI-containing regimen for at least 8 weeks prior to randomization.
6. Patient has on-going viral replication (defined as an HIV-1 viral load of ≥ 500 copies/mL) and a successful virtual phenotype obtained at screening.
7. Any baseline CD4 cell count will be allowed.
8. Karnofsky performance score of ≥ 70.
9. Acceptable screening laboratory values that indicate adequate baseline organ function. Laboratory values are considered acceptable if the following apply:

   * ALT ≤2.5 x ULN and AST ≤2.5 x ULN (≤DAIDS Grade 1, Appendix 10.1).
   * Any DAIDS grade cholesterol, triglycerides, GGT, CPK or LDH is acceptable.
   * All other laboratory test values must be ≤DAIDS Grade 2.
10. Willingness to initiate CD4+ cell count-guided chemoprophylaxis to prevent opportunistic infections.
11. Willingness to abstain from ingesting substances which may alter plasma study drug levels by interaction with the cytochrome P450 system during the study.

Inclusion Criteria:

1. Previous use of Tipranavir (TPV) or Darunavir (DRV).
2. Full genotypic resistance (reported as minimal response) to Tipranavir (TPV) or Darunavir (DRV) on screening virtual phenotype:
3. Female patient of child-bearing potential who:

   has a positive serum pregnancy test at screening, is breast feeding, is planning to become pregnant, is not willing to use double-barrier methods (simultaneous use of two different methods such as diaphragm with spermicidal substance and condom) of contraception or requires ethinyl estradiol administration. Barrier methods of contraception include diaphragm with spermicidal substance, condom for females, cervical caps and condoms.
4. History of Progressive Multifocal Leukoencephalopathy (PML), Visceral Kaposi's Sarcoma (KS), and/or any malignancy.
5. Any AIDS defining illness that is unresolved, symptomatic or not stable on treatment for at least 12 weeks at screening visit.
6. Use of immunomodulatory drugs (such as interferon, cyclosporin, hydroxyurea and interleukin 2) within 30 days prior to randomization.
7. Current use of systemic cytotoxic chemotherapy.
8. All contraindications listed in the product monographs of Aptivus, Prezista and Norvir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (54):
- United States (9):
  - 1182.71.1109 Boehringer Ingelheim Investigational Site, Beverly Hills, California
  - 1182.71.1101 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1182.71.1104 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1182.71.1115 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1182.71.1108 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1182.71.1126 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1182.71.1124 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1182.71.1116 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1182.71.1118 Boehringer Ingelheim Investigational Site, Longview, Texas
- Belgium (4):
  - 1182.71.3202 Boehringer Ingelheim Investigational Site, Brussels
  - 1182.71.3203 Boehringer Ingelheim Investigational Site, Brussels
  - 1182.71.3205 Boehringer Ingelheim Investigational Site, Brussels
  - 1182.71.3206 Boehringer Ingelheim Investigational Site, Charleroi
- Canada (5):
  - 1182.71.1002 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1182.71.1001 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1182.71.1003 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1182.71.1006 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1182.71.1010 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- France (7):
  - 1182.71.3305A Boehringer Ingelheim Investigational Site, Bondy
  - 1182.71.3303A Boehringer Ingelheim Investigational Site, Garches
  - 1182.71.3301A Boehringer Ingelheim Investigational Site, Lyon
  - 1182.71.3312A Boehringer Ingelheim Investigational Site, Lyon
  - 1182.71.3306A Boehringer Ingelheim Investigational Site, Paris
  - 1182.71.3308A Boehringer Ingelheim Investigational Site, Paris
  - 1182.71.3310A Boehringer Ingelheim Investigational Site, Tourcoing
- Germany (3):
  - 1182.71.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 1182.71.4907 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1182.71.4903 Boehringer Ingelheim Investigational Site, Mainz
- Greece (3):
  - 1182.71.3002 Boehringer Ingelheim Investigational Site, Athens
  - 1182.71.3003 Boehringer Ingelheim Investigational Site, Athens
  - 1182.71.3001 Boehringer Ingelheim Investigational Site, Piraeus
- Italy (6):
  - 1182.71.3912 Boehringer Ingelheim Investigational Site, Antella (fi)
  - 1182.71.3901 Boehringer Ingelheim Investigational Site, Brescia
  - 1182.71.3908 Boehringer Ingelheim Investigational Site, Florence
  - 1182.71.3916 Boehringer Ingelheim Investigational Site, Palermo
  - 1182.71.3907 Boehringer Ingelheim Investigational Site, Pavia
  - 1182.71.3919 Boehringer Ingelheim Investigational Site, Pescara
- Portugal (3):
  - 1182.71.3502 Boehringer Ingelheim Investigational Site, Amadora
  - 1182.71.3504 Boehringer Ingelheim Investigational Site, Lisbon
  - 1182.71.3503 Boehringer Ingelheim Investigational Site, Porto
- 1182.71.1129 Boehringer Ingelheim Investigational Site, Ponce, Puerto Rico
- Spain (6):
  - 1182.71.3401 Boehringer Ingelheim Investigational Site, Barcelona
  - 1182.71.3402 Boehringer Ingelheim Investigational Site, Barcelona
  - 1182.71.3403 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1182.71.3405 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.71.3407 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.71.3408 Boehringer Ingelheim Investigational Site, Santiago de Compostela
- Thailand (6):
  - 1182.71.6604 Boehringer Ingelheim Investigational Site, Bangkok
  - 1182.71.6601 Boehringer Ingelheim Investigational Site, Bangkok Noi
  - 1182.71.6605 Boehringer Ingelheim Investigational Site, Chiang Mai
  - 1182.71.6602 Boehringer Ingelheim Investigational Site, Khon Kaen
  - 1182.71.6606 Boehringer Ingelheim Investigational Site, Nonthaburi
  - 1182.71.6603 Boehringer Ingelheim Investigational Site, Phathumwan
- 1182.71.1016 Boehringer Ingelheim Investigational Site, Nassau, The Bahamas

REFERENCES:
- [Derived] Elgadi MM, Piliero PJ. Boosted tipranavir versus darunavir in treatment-experienced patients: observational data from the randomized POTENT trial. Drugs R D. 2011 Dec 1;11(4):295-302. doi: 10.2165/11596340-000000000-00000. PMID 22007990

RESULTS

PARTICIPANT FLOW:
Groups:
- Tipranavir 500 mg/Ritonavir 200 mg: Tipranavir (TPV) 250 mg soft gelatin capsules Ritonavir (RTV) 100 mg soft gelatin capsules dose: 500 mg TPV/200 mg RTV, twice daily mode of admin.: Oral
- Darunavir 600 mg/Ritonavir 100 mg: Prezista® (DRV) 300 mg tablets Ritonavir (RTV) 100 mg soft gelatin capsules dose: 600 mg DRV/100 mg RTV, twice daily mode of admin.: Oral
Period: Overall Study
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Started | 19 | 20
Completed | 0 | 0
Not Completed | 19 | 20
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Early termination of the trial | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.3 (6.1) | 43.1 (6.2) | 43.6 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Time to Virologic Failure Through 48 Weeks of Treatment, Using Viral Load (VL) < 50 Copies/Millilitre (mL) as the Response Criterion.
Time Frame: 48 weeks of treatment
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Treatment Response at Week 48, Using VL < 50 Copies/mL as the Response Criterion and the FDA Definition for Handling Drug Discontinuations ((NCF) Non-Completers=Failure).
Time Frame: 48 weeks of treatment
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Intent-To-Treat Analysis of Virologic Response at Week 48, Using VL < 50 Copies/mL as the Response Criterion Where Patients Are Followed Until Week 48 for VL Regardless of Whether or Not They Remain on Study Drug.
Time Frame: 48 weeks of treatment
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Virologic Failure Through 48 Weeks of Treatment, Using VL < 400 Copies/mL as the Response Criterion.
Time Frame: 48 weeks of treatment
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Response up to 48 Weeks Using VL < 50 Copies/mL Using Censored
Time Frame: up to 48 weeks
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Response up to 48 Weeks Using VL < 50 Copies/mL Using NCF
Time Frame: up to 48 weeks
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Response up to 48 Weeks Using VL < 50 Copies/mL Using Intent-to-treat
Time Frame: up to 48 weeks
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Response up to 48 Weeks Using VL < 400 Copies/mL Using Censored
Time Frame: up to 48 weeks
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Response up to 48 Weeks Using VL < 400 Copies/mL Using NCF
Time Frame: up to 48 weeks
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Response up to 48 Weeks Using VL < 400 Copies/mL Using Intent-to-treat
Time Frame: up to 48 weeks
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Response up to 48 Weeks Using at Least a 1 log10 Reduction in Viral Load From Baseline Using Censored
Time Frame: up to 48 weeks
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Response up to 48 Weeks Using at Least a 1 log10 Reduction in Viral Load From Baseline Using NCF
Time Frame: up to 48 weeks
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Response up to 48 Weeks Using at Least a 1 log10 Reduction in Viral Load From Baseline Using Intent-to-treat
Time Frame: up to 48 weeks
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Daily Average in CD4+ Cell Count Change From Baseline at up to Week 8
Time Frame: up to week 8
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Daily Average in CD4+ Cell Count Change From Baseline up to Week 24
Time Frame: up to week 24
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Daily Average in CD4+ Cell Count Change From Baseline up to Week 48
Time Frame: up to week 48
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Daily Average in Viral Load Change From Baseline up to Week 8
Time Frame: up to week 8
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Daily Average in Viral Load Change From Baseline up to Week 24
Time Frame: up to week 24
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Daily Average in Viral Load Change From Baseline up to Week 48
Time Frame: up to week 48
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change From Baseline in CD4+ Cell Count up to Week 48
Time Frame: up to week 48
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Change From Baseline in log10 Viral Load up to Week 48
Time Frame: up to week 48
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Occurrence of New AIDS Progression Events or Death
Time Frame: through 48 weeks of treatment
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent onwards through the observational phase (50 weeks).
Arm/Group | Tipranavir 500 mg/Ritonavir 200 mg | Darunavir 600 mg/Ritonavir 100 mg
Serious Adverse Events (participants affected / at risk) | 0/19 | 2/20
Other Adverse Events (participants affected / at risk) | 12/19 | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tipranavir 500 mg/Ritonavir 200 mg (N=19) | Darunavir 600 mg/Ritonavir 100 mg (N=20)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Iliac artery thrombosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tipranavir 500 mg/Ritonavir 200 mg (N=19) | Darunavir 600 mg/Ritonavir 100 mg (N=20)
Angina pectoris (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 1 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Pyrexia (General disorders) | 0 | 2
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Facial wasting (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.